CLINICAL TRIAL: NCT04328701
Title: Prediction of Outcomes Following Total Knee Replacement- Pilot
Acronym: POKR-p
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Robert Edwards, Clinical Psychologist, Brigham and Women's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2010P000978-p
Record Dates: First submitted 2020-02-03; First posted 2020-03-31 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Osteoarthritis, Knee; Knee Replacement
Keywords: CBT
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: All participants will undergo quantitative sensory testing, physical functioning testing, and pain-related outcomes assessment. Participants in the intervention arm will undergo brief mindfulness-based cognitive behavioral sessions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-based CBT (Experimental): All participants will receive four individual mindfulness-based CBT sessions.
  Interventions: Behavioral: Mindfulness-based Cognitive Behavioral Therapy
- Treatment as Usual (No Intervention): All participants will undergo surgery as usual, with no additional intervention.

INTERVENTIONS:
Behavioral: Mindfulness-based Cognitive Behavioral Therapy — Mindfulness-based CBT methods are based on pain self-management paradigms, and involve the identification and reduction of maladaptive pain-related cognitions (i.e., catastrophizing), the enhancement of self-efficacy for managing pain, and training in the use of adaptive pain-coping strategies such as relaxation, distraction, and self-talk.
  Arms: Mindfulness-based CBT

SUMMARY:
This study seeks to examine multiple risk factors as predictors of pain and function following total knee arthroplasty (TKA). Risk factors will be measured pre-surgically using psychophysical testing procedures, multimodal evaluation of sleep, standardized questionnaires. Additionally, this study will collect pilot data on a brief mindfulness-based cognitive-behavioral treatment that may help to improve long-term TKA outcomes.

The pilot study compared TKA patients that received brief mindfulness-based cognitive behavioral therapy (MBCBT) to the treatment-as-usual (TAU) group from the parent study.

DETAILED DESCRIPTION:
The present study seeks to collect pilot data on a brief mindfulness-based cognitive-behavioral treatment to determine the feasibility of this intervention and its potential benefits. The study includes 6 total contacts, 1 visit before surgery and 3 after surgery, and 2 phone calls. The last visit will be about 6 months after surgery. The study includes evaluation of peoples' pain, physical functioning, medication use, and physiological responses to sensory stimuli such as heat and cold. The research takes place at the Brigham & Women's Pain Management Center, 850 Boylston St, Chestnut Hill.

ELIGIBILITY:
Inclusion Criteria:

1. Age 45 or older,
2. Meet the American College of Rheumatology criteria for knee OA,
3. Scheduled to undergo total knee arthroplasty,
4. Facility with the English language that is adequate to complete study procedures

Exclusion Criteria:

1. Cognitive impairment preventing completion of study assessment procedures.
2. Myocardial infarction within the past 12 months.
3. Presence of Severe Raynaud's or severe neuropathy,
4. Active vasculitis or severe peripheral vascular disease,
5. Current infection,
6. Use of oral steroids,
7. Recent history of substance abuse or dependence,
8. Known anemia

Ages: 45 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Brief Pain Inventory (BPI) | baseline
  Measure of pain severity and pain interference
Brief Pain Inventory (BPI) | 6-week
  Measure of pain severity and pain interference
Brief Pain Inventory (BPI) | 3-months
  Measure of pain severity and pain interference
Brief Pain Inventory (BPI) | 6-months
  Measure of pain severity and pain interference

SECONDARY OUTCOMES:
Quantitative Sensory Testing (QST) | baseline
  Measures of responses to standardized stimuli
Quantitative Sensory Testing (QST) | 3-months
  Measures of responses to standardized stimuli
Pain Catastrophizing Scale | baseline
  Assess catastrophic thinking related to pain
Pain Catastrophizing Scale | 6-week
  Assess catastrophic thinking related to pain
Pain Catastrophizing Scale | 3-months
  Assess catastrophic thinking related to pain
Pain Catastrophizing Scale | 6-months
  Assess catastrophic thinking related to pain
PROMIS-SF | baseline
  Measures anxiety and depression symptoms
PROMIS-SF | 6-week
  Measures anxiety and depression symptoms
PROMIS-SF | 3-months
  Measures anxiety and depression symptoms
PROMIS-SF | 6-months
  Measures anxiety and depression symptoms
The Western Ontario McMaster Universities Osteoarthritis Scale (WOMAC) | baseline
  24 items and is a well-validated, widely-used outcomes measure that yields three indices specific to osteoarthritis: 1) pain, 2) disability and 3) joint stiffness, which are sensitive to treatment, with internal consistency coefficients for all scales above 0.8.
The Western Ontario McMaster Universities Osteoarthritis Scale (WOMAC) | 6-week
  24 items and is a well-validated, widely-used outcomes measure that yields three indices specific to osteoarthritis: 1) pain, 2) disability and 3) joint stiffness, which are sensitive to treatment, with internal consistency coefficients for all scales above 0.8.
The Western Ontario McMaster Universities Osteoarthritis Scale (WOMAC) | 3-months
  24 items and is a well-validated, widely-used outcomes measure that yields three indices specific to osteoarthritis: 1) pain, 2) disability and 3) joint stiffness, which are sensitive to treatment, with internal consistency coefficients for all scales above 0.8.
The Western Ontario McMaster Universities Osteoarthritis Scale (WOMAC) | 6-months
  24 items and is a well-validated, widely-used outcomes measure that yields three indices specific to osteoarthritis: 1) pain, 2) disability and 3) joint stiffness, which are sensitive to treatment, with internal consistency coefficients for all scales above 0.8.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Edwards, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital Pain Management Center, Chestnut Hill, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pester BD, Wilson JM, Yoon J, Lazaridou A, Schreiber KL, Cornelius M, Campbell CM, Smith MT, Haythornthwaite JA, Edwards RR, Meints SM. Brief Mindfulness-Based Cognitive Behavioral Therapy is Associated with Faster Recovery in Patients Undergoing Total Knee Arthroplasty: A Pilot Clinical Trial. Pain Med. 2023 Jun 1;24(6):576-585. doi: 10.1093/pm/pnac183. PMID 36394250
- See also: Local site recruitment link — https://rally.partners.org/study/knee_replacement